CLINICAL TRIAL: NCT00667914
Title: A New Clinical Pathway for Patients With Fractured Neck of Femur - The Orthopedics Operate, the Geriatricians Manage the Medical Work-up
Brief Title: A New Clinical Pathway for Patients With Fractured Neck of Femur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2008.335 (REC)
Record Dates: First submitted 2008-04-18; First posted 2008-04-28 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Hip Fracture; Aged
Keywords: Hip-unit; Geriatric care; Mobility; Site of residence
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthogeriatric unit (Experimental): Geriatric work-up on hip-fracture patients
  Interventions: Procedure: geriatric work-up
- Orthopedic care as usual (Active Comparator): Traditional care in the orthopedic unit
  Interventions: Procedure: Orthopedic care as usual

INTERVENTIONS:
Procedure: geriatric work-up — Pre- and postoperative treatment of hip-fracture patients in an orthogeriatric unit(geriatric evaluation and management)
  Other Names: Geriatric work-up in hip-fracture patients
  Arms: Orthogeriatric unit
Procedure: Orthopedic care as usual — treatment in ordinary orthopedic unit
  Arms: Orthopedic care as usual

SUMMARY:
The intention is to evaluate the effectiveness of a multi-factorial medical treatment of patients with hip fractures in a specially designed unit for elderly hip fracture patients (orthogeriatric unit) as compared to traditional care in an orthopedic unit.

DETAILED DESCRIPTION:
The intention of the present project is to evaluate the effectiveness of multi-factorial medical treatment of patients with hip fractures in a specially designed geriatric unit for elderly hip fracture patients (orthogeriatric unit) as compared to traditional care in an orthopedic unit.

Every year 9000 patients undergo surgery for hip fractures in Norway. The epidemic of hip fractures is among the most common causes of acute hospitalization of older people and is associated with high morbidity, mortality, disability and subsequent hospital and social costs as well as reduction in quality of life.

Traditionally hip fracture surgery is performed and followed by care in orthopedic departments. Additional rehabilitation within the hospital is sometimes provided by a geriatrician and a team of rehabilitation specialists, but there is a lot of variety in these rehabilitation programmes. Studies have shown improved outcomes when older people were cared for by a specialist multidisciplinary team. However, the results are not conclusive and more research is needed also in that field, as stated by a Cochrane review.

It is well known that hip-fracture patients are frequently characterized by high age, co-morbidity and frailty, which may often be the main reason for falls and injuries as hip fractures. In a previous project performed by our group we showed that by treating acutely sick, frail elderly patients in a geriatric evaluation and management unit mortality was significantly reduced and patients' chances of living at home was improved. Later our research group has focused on assessment and treatment of older persons at risk of falling. Now we have started to focusing on the ultimate consequence of falling in frail elderly people: the hip fracture, through an observational study. The present study is partly also a consequence of this.

The present project will primarily examine the effect of establishing a radical and new clinical pathway for patients with hip fracture starting immediately at admittance to hospital by randomizing patients to treatment in an orthogeriatric unit (intervention group) or to treatment in orthopedic wards (control group) in the emergency department. There will be no specific follow-up after discharge from hospital.

Primary endpoints will evaluate possible effects on mobility as measured by Short Physical Performance Battery (SPPB). As secondary endpoints other relevant functional aspects, site of residence, health economic variables and mortality will be studied. This study will give increased scientific understanding of whether treatment in a specialized orthogeriatric unit can improve outcomes as mobility, the extensive numbers of nursing home admissions and high mortality after a hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* age >70 years
* living in nearby municipalities
* able to walk 10 m before fracture
* medial, pertrochanteric and subtrochanteric hip-fractures

Exclusion Criteria:

* nursing home residents
* expected to die within 3 months
* pathological fractures

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 397 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mobility | 1, 4 and 12 months after surgery

SECONDARY OUTCOMES:
Site of residence | 1, 4 and 12 months after surgery
Other functional aspects than mobility | 1, 4 and 12 months after surgery
Health economic variables | 1, 4 and 12 months after surgery
Mortality | 1, 4 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olav Sletvold, MD. Ph D, Principal Investigator — Department of Neuroscience, Norwegian University of Science and Technology

REFERENCES:
- [Background] Sletvold O, Helbostad JL, Thingstad P, Taraldsen K, Prestmo A, Lamb SE, Aamodt A, Johnsen R, Magnussen J, Saltvedt I. Effect of in-hospital comprehensive geriatric assessment (CGA) in older people with hip fracture. The protocol of the Trondheim Hip Fracture trial. BMC Geriatr. 2011 Apr 21;11:18. doi: 10.1186/1471-2318-11-18. PMID 21510886
- [Background] Prestmo A, Saltvedt I, Helbostad JL, Taraldsen K, Thingstad P, Lydersen S, Sletvold O. Who benefits from orthogeriatric treatment? Results from the Trondheim hip-fracture trial. BMC Geriatr. 2016 Feb 19;16:49. doi: 10.1186/s12877-016-0218-1. PMID 26895846
- [Result] Prestmo A, Hagen G, Sletvold O, Helbostad JL, Thingstad P, Taraldsen K, Lydersen S, Halsteinli V, Saltnes T, Lamb SE, Johnsen LG, Saltvedt I. Comprehensive geriatric care for patients with hip fractures: a prospective, randomised, controlled trial. Lancet. 2015 Apr 25;385(9978):1623-33. doi: 10.1016/S0140-6736(14)62409-0. Epub 2015 Feb 5. PMID 25662415
- [Result] Taraldsen K, Thingstad P, Sletvold O, Saltvedt I, Lydersen S, Granat MH, Chastin S, Helbostad JL. The long-term effect of being treated in a geriatric ward compared to an orthopaedic ward on six measures of free-living physical behavior 4 and 12 months after a hip fracture - a randomised controlled trial. BMC Geriatr. 2015 Dec 4;15:160. doi: 10.1186/s12877-015-0153-6. PMID 26637222
- [Result] Haugan K, Johnsen LG, Basso T, Foss OA. Mortality and readmission following hip fracture surgery: a retrospective study comparing conventional and fast-track care. BMJ Open. 2017 Aug 29;7(8):e015574. doi: 10.1136/bmjopen-2016-015574. PMID 28851773
- [Result] Thingstad P, Taraldsen K, Saltvedt I, Sletvold O, Vereijken B, Lamb SE, Helbostad JL. The long-term effect of comprehensive geriatric care on gait after hip fracture: the Trondheim Hip Fracture Trial--a randomised controlled trial. Osteoporos Int. 2016 Mar;27(3):933-942. doi: 10.1007/s00198-015-3313-9. Epub 2015 Sep 14. PMID 26370827
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Taraldsen K, Sletvold O, Thingstad P, Saltvedt I, Granat MH, Lydersen S, Helbostad JL. Physical behavior and function early after hip fracture surgery in patients receiving comprehensive geriatric care or orthopedic care--a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2014 Mar;69(3):338-45. doi: 10.1093/gerona/glt097. Epub 2013 Jul 31. PMID 23902933